CLINICAL TRIAL: NCT01272414
Title: Use of Botox in the Management of Thyroid Related Upper Eyelid Retraction
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: lack of funding
Sponsor: University of Toronto (Other)
Collaborators: Allergan (Industry)
Responsible Party: Dr Nancy Tucker, MD FRCSC, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-0261-A
Record Dates: First submitted 2011-01-06; First posted 2011-01-07 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2010-12

CONDITIONS: Graves Ophthalmopathy
Keywords: Eyelid retraction; Botulinum Toxins
MeSH Terms: conditions — Graves Ophthalmopathy | interventions — Botulinum Toxins, Type A; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- BoTox Treatment (Experimental): Subjects receive BoTox injection to levator complex
  Interventions: Drug: Botulinum Toxin Type A
- Saline injection (Placebo Comparator): Saline injection to levator complex
  Interventions: Drug: Saline injection

INTERVENTIONS:
Drug: Botulinum Toxin Type A — 2-12 units in weekly 2u doses to effect
  Other Names: BoTox
  Arms: BoTox Treatment
Drug: Saline injection — Injection of 0.4cc 0.9% normal saline
  Other Names: Placebo
  Arms: Saline injection

SUMMARY:
Currently there are few therapeutic options for the treatment of lid retraction secondary to thyroid orbitopathy (TO) during the active stages of the disease. BoTox injection is capable of creating a ptosis, that in the setting of TO can return the upper lid to a more physiologic position, thus improving cosmesis, corneal lubrication and potentially quiescent stage lid position. This investigation aims to examine the properties of this relationship.

ELIGIBILITY:
Inclusion Criteria:

* Active stage thyroid orbitopathy, as determined by symptom onset of under 6 months.
* Upper eyelid retraction of 1mm or greater.
* Complaining of either significant ocular symptoms (despite appropriate use of ocular lubricants), or bothered by the cosmetic deformity associated with the eyelid retraction.

Exclusion Criteria:

* Less than 18 years of age
* Age over 65 years
* Pregnant or nursing
* Known peripheral neuropathy or neuromuscular junction disorder
* Demonstrated allergy to BoTox
* Current infection over the injection site
* Are currently taking any of the following medications: aminoglycosides, penicillamine, quinine, and calcium channel blockers.
* Previous or concurrent prednisone therapy
* Undergone previous upper eyelid surgery
* Severe vision threatening TO

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Estimated); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction in upper lid retraction (in mm) | 4 month

SECONDARY OUTCOMES:
Subjective improvement in lid retraction related dry eye symptoms | 4 months
  ocular surface disease index score
Subjective improvement in lid retraction related cosmesis | 4 months
  Graves Orbitopathy quality of life score

CONTACTS AND LOCATIONS:
Overall Officials: Daniel B Rootman, MSc MD, Principal Investigator — University of Toronto; Nancy Tucker, MD FRCSC, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada